CLINICAL TRIAL: NCT07266064
Title: Repeated Botulinum Toxin Type A Injections on the Masseter Muscle of Individuals With Sleep Bruxism: A Longitudinal Ultrasonographic Study.
Brief Title: Repeated Botulinum Toxin Type A Injections on Intramuscular Fat Accumulation in Individuals With Sleep Bruxism.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Volkan Yazici (Other)
Responsible Party: Sponsor-Investigator, Melek Volkan Yazici, Associate Professor, Yuksek Ihtisas University
Organization: Yuksek Ihtisas University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Botox series
Record Dates: First submitted 2025-11-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Bruxism; Bruxism, Sleep; Bruxism, Sleep-Related
Keywords: Botulinum Toxin Type A; Bruxism; Masseter Muscle; Ultrasonography; Adipose Tissue; Longitudinal Study
MeSH Terms: conditions — Bruxism; Sleep Bruxism

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal study.
Masking Description: The radiologist who acquired the ultrasonographic data and the researcher who performed the cross-sectional fat infiltration analysis were completely blinded to each other's procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BoNT-A (Experimental): At baseline, all participants underwent ultrasonographic evaluation of both masseter muscles (U0). Two weeks later, the first BoNT-A injection was administered bilaterally (U1). Thereafter, ultrasonography was repeated at six-month intervals (U1-U4). Each of the intermediate assessments was followed by a BoNT-A injection two weeks later (U2-U4), whereas the final assessment (U4) was not followed by injection. Thus, the protocol comprised five ultrasound sessions (U0-U4) and four BoNT-A sessions (U1-U4), unless the participant discontinued the study. All ultrasound examinations were performed by the same experienced examiner using the same device and standardized probe settings.
  Interventions: Other: Botilinum Toxin injection

INTERVENTIONS:
Other: Botilinum Toxin injection — This prospective longitudinal interventional study included adults with probable sleep bruxism who received bilateral BoNT-A injections every six months, with ultrasonographic assessments also performed at six-month intervals, immediately before each new injection. The protocol therefore comprised four injection cycles and five ultrasound sessions. Ultrasonographic evaluations were conducted before the first injection and six months after each subsequent injection to quantify intramuscular fat percentage at rest and during maximum voluntary contraction. Fat area percentage was computed from standardized B-mode images using binary segmentation in CT-Analyzer software.

SUMMARY:
This study investigates whether repeated botulinum toxin type A (BoNT-A) injections used to manage sleep bruxism lead to structural changes-specifically intramuscular fat accumulation-in the masseter muscle. Adults with probable sleep bruxism receive BoNT-A injections every six months and undergo ultrasound evaluations before each injection. By tracking fat percentage in the masseter muscle over multiple treatment cycles, the study aims to determine whether long-term BoNT-A use causes progressive structural alterations or remains safe for repeated clinical use.

DETAILED DESCRIPTION:
Botulinum toxin type A (BoNT-A) is commonly used for the management of sleep bruxism, yet concerns persist regarding its long-term effects on muscle structure, including the possibility of intramuscular fat accumulation in the masseter muscle. This prospective longitudinal study follows adults with probable sleep bruxism who receive bilateral BoNT-A injections at six-month intervals. Ultrasound imaging is performed immediately before each injection, resulting in four injection cycles and five standardized ultrasound assessments.

Intramuscular fat percentage is quantified from B-mode images at rest and during maximum voluntary contraction using binary segmentation techniques. By examining changes over repeated treatment cycles, the study evaluates whether BoNT-A leads to progressive fat infiltration or instead demonstrates a stable or adaptive pattern. Findings will help clarify the structural safety of long-term BoNT-A use in non-spastic masticatory muscles and guide clinical decision-making for ongoing bruxism management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Clinical diagnosis of probable sleep bruxism according to the international consensus criteria proposed by Lobbezoo et al.
* Indication for BoNT-A injection in the masseter muscle due to bruxism-related pain or muscle hypertrophy.
* Willingness to undergo repeated BoNT-A injections at six-month intervals.
* Willingness to participate in ultrasonographic evaluations at each follow-up visit.

Exclusion Criteria:

* Presence of neurological or neuromuscular disorders affecting the masticatory muscles (e.g., dystonia, myasthenia gravis).
* History of orofacial trauma, temporomandibular joint dysfunction, or maxillofacial surgery.
* Systemic diseases that may affect neuromuscular transmission or muscle metabolism.
* Use of medications known to interfere with neuromuscular function, including aminoglycoside antibiotics or corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic imaging | From enrollment to 6 months
  Cross-sectional imaging was obtained from the same anatomical plane. The probe position was determined at each visit using consistent anatomical landmarks-specifically the lower border of the mandibular corpus and the thickest region of the masseter muscle. The imaging plane part of the masseter, located between the posterior border adjacent to the parotid gland and the anterior border of the mandibular ramus. Ultrasonographic images were acquired both at rest (RST) and during maximum voluntary contraction (MVC) under identical device settings by the same experienced radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: GOKHAN YAZICI, A/Prof, Study Chair — Gazi University
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to ethical and confidentiality considerations, the dataset generated and/or analyzed during the current study is not publicly available. However, data may be made available from the corresponding author upon reasonable request and subject to institutional approval.